CLINICAL TRIAL: NCT07310875
Title: Gastric Ultrasound in Patients Who Have Undergone Bariatric Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Malikah Latmore, Regional Anesthesia and Acute Pain Medicine Fellowship Director, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY-23-01595
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Weight Loss; Gastrectomy
Keywords: Point of Care Ultrasound; Sleeve gastrectomy
MeSH Terms: conditions — Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Gastric Point of Care Ultrasound (POCUS) group (Experimental): Participates scheduled to undergo bariatric surgery and have had no prior abdominal surgery.
  Interventions: Procedure: Gastric Point of Care Ultrasound

INTERVENTIONS:
Procedure: Gastric Point of Care Ultrasound — After the patient has undergone intubation, the patient will be positioned in the supine and then the right lateral decubitus position on the operating room table. A curvilinear ultrasound probe with gel will be placed on the patient below the xiphoid process. A picture is then obtained of the antrum of the stomach. The probe may need to be moved, tilted, or rotated to obtain the clearest image of the antrum of the stomach. After the images are obtained, the patient will be repositioned to supine for the procedure. Once the surgical procedure is complete, the patient will once again undergo gastric POCUS prior to extubation.

SUMMARY:
This is a nonrandomized prospective study. The purpose is to describe how to image the stomachs of patients after the patients have had bariatric surgery. Participants will have the stomachs imaged while undergoing general anesthesia for a bariatric procedure pre-operatively and post-operatively using point-of-care ultrasound (POCUS). The pre-operative imaging will be done post-intubation and the post-operative imaging will be done pre-extubation. There are minimal risks to gastric POCUS. Risks typically include discomfort to the patient, which will be avoided as the patient will be under general anesthesia at the time of imaging.

DETAILED DESCRIPTION:
Aspiration of gastric contents in the perioperative period is a well-known complication with potentially disastrous consequences. Gastric POCUS is a tool clinicians can utilize to assess stomach fullness and risk stratify prior to induction of anesthesia. There is currently no literature describing how bariatric surgeries impact the location of the stomach and/or the ability of clinicians to obtain gastric POCUS images. Recent increased use of GLP-1 agonists, which delay gastric emptying, has renewed conversations surrounding using gastric POCUS to assess aspiration risk. Case reports have been published showing aspiration events in patients taking GLP-1 agonists despite an adequate fasting period. Additionally, recent studies have shown that these medications can help patients who have undergone bariatric surgery and then regained the weight, lose said weight. Given the possibility that patients may be post-bariatric surgery and currently taking GLP-1 agonists, POCUS is an important skill to utilize that can help anesthesiologists assess aspiration risk. This study will aim to fill a gap in the literature by describing how bariatric surgery can impact the location of the stomach and how to obtain sonographic images of the stomach in a post-bariatric surgery abdomen. The analysis will include description of how the images were obtained (ex: needing to rotate the probe further than expected, or stomach displacement, etc.) and comparison to the procedure used to obtain preoperative images. The measurements will be subjective to the PI who is certified in POCUS use.

Discussions will be held with surgeons who perform bariatric surgery, to determine which patients fit the qualifications to participate in the study. Patients are routinely seen by anesthesiologists for their anesthetic evaluation in the pre-operative holding area on the day of their procedure. After the patient have been evaluated, the patient will have time to discuss the study with the anesthesia team prior to transferring the patient to the OR. Consent will be obtained in the preoperative holding area. There are sequestered rooms in this area where patients can be brought for increased privacy during the consent process. The team will finalize participation and ask the participant to sign the study consent forms. All patient will be provided with copies of the IRB protocol and consent if the patient wish to have it. If agreeable to joining the study, the patient will undergo gastric POCUS after intubation. To perform the gastric POCUS, the patient will be in the supine position and the right lateral decubitus position on the operating room table. A curvilinear ultrasound probe with gel will be placed on the patient just below the xiphoid. A picture is then obtained of the antrum of the stomach. The probe may need to be moved, tilted, or rotated to obtain the clearest image of the antrum of the stomach. The POCUS of the abdomen before abdominal surgery will be done before the surgical team has prepared a sterile field for their surgery. Therefore, there is no need to maintain sterile precautions when using the ultrasound on the abdomen. Once the surgical procedure is complete, the patient will once again undergo gastric POCUS before extubation.

ELIGIBILITY:
Inclusion Criteria:

* 18-85 years old
* scheduled to undergo bariatric surgery
* no prior abdominal surgery

Exclusion Criteria:

* ASA physical status > 3
* Urgent or emergent surgery
* Patient refusal or inability to consent
* Prior abdominal surgery

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in distance from peritoneal wall | end of the individual's procedure, at 2 hrs after procedure start on postoperative day 0
  Range: 3-5 cm. Higher score indicates greater displacement and less utility of gastric point-of-care ultrasound in these patients.
Gastric antrum Cross-sectional area (CSA) | end of the individual's procedure, at 2 hrs after procedure start
  Range: 1-10 centimeters squared. Gastric antrum Cross-sectional area (CSA) is a calculated product of Anteroposterior (AP) Diameter and Craniocaudal (CC) diameter. (CSA = AP x CC) Higher score means that patient has a larger gastric volume and is at a higher aspiration risk.

SECONDARY OUTCOMES:
Anteroposterior (AP) Diameter | end of the individual's procedure, at 2 hrs after procedure start
  Range: 0-10 centimeters. Higher score means that patient has a larger gastric volume and is at a higher aspiration risk.
Craniocaudal (CC) diameter | end of the individual's procedure, at 2 hrs after procedure start
  Range: 0-10 centimeters. Higher score means that patient has a larger gastric volume and is at a higher aspiration risk.
Postoperative aspiration events | until day of hospital discharge, average 1-3 days
  Number of Postoperative aspiration events

CONTACTS AND LOCATIONS:
Overall Officials: Malikah Latmore, MD, Principal Investigator — Mount Sinai Morningside Hospital
Locations (1):
- Mount Sinai West and Morningside, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ('learned intermediary') identified for this purpose.
  To achieve aims in the approved proposal. Proposals should be directed to Malikah.Latmore@mountsinai.org. To gain access, data requestors will need to sign a data access agreement. Data are available for 5 years at a third party website (Link tbd).

REFERENCES:
- [Background] Pai SL, Bojaxhi E, Logvinov II, Porter SB, Feinglass NG, Robards CB, Torp KD. Ultrasound Assessment of Gastric Volume After Bariatric Surgery: A Case Report. A A Pract. 2019 Jan 1;12(1):1-4. doi: 10.1213/XAA.0000000000000824. PMID 29985844
- [Background] Smith G, Ng A. Gastric reflux and pulmonary aspiration in anaesthesia. Minerva Anestesiol. 2003 May;69(5):402-6. PMID 12768174
- [Background] Gulak MA, Murphy P. Regurgitation under anesthesia in a fasted patient prescribed semaglutide for weight loss: a case report. Can J Anaesth. 2023 Aug;70(8):1397-1400. doi: 10.1007/s12630-023-02521-3. Epub 2023 Jun 6. PMID 37280458